CLINICAL TRIAL: NCT00373022
Title: The Effect of Moderate Physical Activity on the Physical and Emotional Recovery of Patients With a History of Colorectal Cancer
Brief Title: Moderate Physical Activity in Helping Patients Recover Physically and Emotionally From Stage II Or Stage III Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ana Maria Lopez, MD, Arizona Cancer Center at University of Arizona Health Science Center
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000491199; P30CA023074 (NIH); UARIZ-A04.04
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2006-12

CONDITIONS: Anxiety Disorder; Colorectal Cancer; Depression; Psychosocial Effects of Cancer and Its Treatment
Keywords: depression; anxiety disorder; psychosocial effects of cancer and its treatment; stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Anxiety Disorders; Colorectal Neoplasms; Depression; Colonic Neoplasms; Rectal Neoplasms | interventions — Flow Cytometry; Psychiatric Rehabilitation

INTERVENTIONS:
Behavioral: exercise intervention
Other: flow cytometry
Other: laboratory biomarker analysis
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Physical activity may prevent or lessen depression and anxiety and improve quality of life and immune function in patients with colorectal cancer.

PURPOSE: This randomized clinical trial is studying how well physical activity helps patients with stage II or stage III colorectal cancer recover from cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the effect of moderate physical activity interventions in ameliorating quality of life (as measured by the Functional Assessment of Cancer Therapy-Colon questionnaire) in patients undergoing or who have previously received chemotherapy for stage II or III colorectal cancer.

Secondary

* Assess the effect of different moderate physical activity interventions in ameliorating depression (as measured by the Beck Depression Inventory) and anxiety (as measured by the Spielberger State-Trait Anxiety Inventory) in these patients.
* Assess the effect of these interventions on attitudes related to physical activity (as measured by the American Council on Exercise History questionnaire) in these patients.
* Characterize serum levels and patterns of immune function (cytokines, neutrophils, T cells, B cells, natural killer [NK] cells, and immunoglobulin) in these patients.
* Correlate serum levels and patterns of immune function (cytokines, neutrophils, T cells, B cells, NK cells, and immunoglobulin) with the patients' physical activity levels.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients participate in individual walking sessions once a week for 8 weeks. The sessions include a fitness-related discussion, warm-up and stretch, 45 minutes of physical activity consisting of walking (progressing in intensity), and a cool-down period.
* Arm II: Patients participate in a group walking sessions once a week for 8 weeks. The sessions include a fitness-related discussion, warm-up and stretch, 45 minutes of physical activity consisting of walking (progressing in intensity as in arm I), and a cool-down period.
* Arm III: Patients participate in self-directed physical activity sessions (1½ hours) once a week for 8 weeks. The sessions include warm-up and stretch followed by 45 minutes of progressively intensified physical activity that integrates fundamentals of movement, dance, and exercise principles from established movement methods (i.e., yoga) and a relaxation session/cool-down period.

All patients complete self-reported questionnaires (Spielberger State-Trait Anxiety Inventory, Beck Depression Inventory, Functional Assessment of Cancer Therapy-Colon, and American Council on Exercise History questionnaires). Patients also undergo blood collection at baseline, at 4 weeks, upon completion of study treatment, and at 4 months after completion of study treatment for correlative studies. Blood is examined by flow cytometry for immune function and cytokines.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage II-III colorectal cancer meeting 1 of the following criteria:

  * Undergoing concurrent chemotherapy
  * Completed chemotherapy within the past 2 years

PATIENT CHARACTERISTICS:

* No physical or emotional impairment that would limit study compliance
* No prior or current chronic substance abuse

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Effect of moderate physical activity on quality of life as measured by the Functional Assessment of Cancer Therapy-Colon questionnaire

SECONDARY OUTCOMES:
Effect of moderate physical activity on depression and anxiety as measured by the Beck Depression Inventory and the Spielberger State-Trait Anxiety Inventory
Effect of moderate physical activity on attitudes related to physical activity as measured by the American Council on Exercise History questionnaire
Serum levels and patterns of immune function as measured by cytokine, neutrophil, T cell, B cell, natural killer (NK) cell, and immunoglobulin levels
Correlation of serum levels and patterns of immune function (cytokine, neutrophil, T cell, B cell, NK cell, and immunoglobulin levels) with physical activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Lopez, MD, MPH, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States